CLINICAL TRIAL: NCT07251478
Title: Transparent Communication to Improve Mental Wellbeing and Public Attitude Towards the Reintegration of Former Boko Haram Members in Nigeria: A Pilot Randomised Control Trial
Brief Title: Transparent Communication to Improve Mental Wellbeing and Attitude Towards Reintegration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: Jos University Teaching Hospital (Other); University of Manchester (Other)
Responsible Party: Principal Investigator, Tarela Ike, Senior Lecturer and Principal Investigator, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313g
Record Dates: First submitted 2025-05-20; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety; Trauma; Stress; Trauma, Psychological
Keywords: Anxiety; Depression; Reintegration; Trauma
MeSH Terms: conditions — Depression; Anxiety Disorders; Wounds and Injuries; Psychological Trauma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE) (Experimental): The Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE) intervention is a low-intensity intervention lasting 3-5 minutes.
  Interventions: Behavioral: Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE)
- Control - Waitlist Group (No Intervention): The control group will not receive an intervention until after the assessment periods at baseline (day 1), and end of intervention (day 2) before they will be administered the PEACE intervention.

INTERVENTIONS:
Behavioral: Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE) — The Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE) intervention is a low-intensity intervention lasting 3-5 minutes. The intervention is underpinned by awareness creation, reducing depression and anxiety and the purpose of reintegration programme to encourage change in negative attitudes towards reintegration. The recorded message introduction will commence with a welcome address on the topic, and this is followed by the core message and a closing remark. The core message is composed of three key ambits: 1) emphasizing mental health and welbeing alongside the importance of the reintegration programme, the rationale behind the reintegration programme, including the provision of incentives to dissuade reoffending, (ii) the need for empathy, prosociality, and positive social identity and advantages of reintegration and (iii) calling on the public to forgive and accept them back. The programme will end with a thank you to the audience for listening.
  Arms: Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE)

SUMMARY:
Reintegrating those once affiliated with proscribed terrorist groups constitutes significant global challenges due to public stigma, poor awareness of reintegration programmes and resentment towards incentives provided to rehabilitated former members of such groups. Of central concern is the anxiety, trauma and depression suffered alongside distrust for reintegration programmes, including the genuine repentance of former members of the proscribed group. The implication is its risk in exacerbating reoffending. Yet, a gap exists to address this urgent problem. The proposed study seeks to test and pilot the feasibility and acceptability of a novel intervention called Prosociality, Empathy and Awareness Communication to aid rEintegration (PEACE) in improving mental well-being and public attitude towards reintegration. The intervention is a low-intensity intervention lasting approximately 3-5 minutes design to create awareness on the rationale behind reintegration programme, reduce anxiety, depression and foster positive attitude towards reintegration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Able to provide full consent for their participation.
* A resident of the study areas

Exclusion Criteria:

* Less than 18 years
* Unable to consent
* Currently undergoing severe mental health treatment
* Unable to speak the English language fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Service Satisfaction Scale | At the end of intervention (day 2)
  A five item scale that can be used to assess and measure satisfaction, acceptability and quality of the intervention. Higher score denote positive outcomes and acceptability. Lower score denotes poor satisfaction and acceptability.

SECONDARY OUTCOMES:
Post-traumatic Stress Disorder Checklist (PCL-5) | Baseline (day 1) and at the end of intervention (day 2)
  The PCL-5 is a 20-item self-report measure that can be used to assess the 20 DSM-5 symptoms of post traumatic stress disorder. A 5-10 point change represents reliable change (i.e., change not due to chance) and a 10-20 point change represents clinically significant change.
Generalised Anxiety Disorder (GAD-7) | Baseline (day 1) and at the end of intervention (day 2)
  The GAD-7 is a seven item scale for screening, measuring and assessing the severity of generalised anxiety disorder. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Oslo Social Support Scale (OSSS-3) | Baseline (day 1) and at the end of intervention (day 2)
  The scale is a 3-item self-reported measure designed for assessing and measuring the level of social support. The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support as indicated as follows: a) 3-8 poor social support, b) 9-11 moderate social support, c) 12-14 strong social support.
Patient Health Questionnaire (PHQ-9) | Baseline (day 1) and at the end of intervention (day 2)
  The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that will be used for screening, monitoring, measuring and assessing the severity of depression. Low scores (e.g. 0-4) indicate no depression, however, higher scores (20-27) indicates severe depression.
European Quality of Life Scale EQ-5D-5L | Baseline (day 1) and at the end of intervention (day 2)
  The EQ-5D-5L is a 5 item scale designed to aid assessment of the generic quality of life. In the EQ-5D-5L, each dimension has five response levels: no problems (Level 1); slight (Level 2); moderate (Level 3); severe (Level 4); and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Legal-informed Awareness of Complaint Channel Scale (LACCS) | Baseline (day 1) and at the end of intervention (day 2)
  The LACCS is a 10-item scale that is designed for assessing and measuring level of awareness of complaint channels and legal rights. The scale has an overall rating of 30, with 0-7 indicating poor knowledge, 8-15 (average knowledge), 16-22 (good knowledge) and 23-30 (excellent knowledge).
Attitude Towards Repentant Terrorist and their Reintegration Scale (ATRTRS) | Baseline (day 1) and at the end of intervention (day 2)
  The scale os a 26-item scale that is designed for assessing attitude towards repentant terrorist and their reintegration. The scale has a total score of 130 and assigned the following rating: 1 = Extremely poor reintegration attitude (1-26); 2 = Poor reintegration attitude (27-52); 3 = Moderate attitude towards reintegration (53-78); 4 = Good attitude towards reintegration (79-104); and 5 = Very good attitude towards reintegration (105-130).

OTHER OUTCOMES:
Vignette | Baseline (day 1) and at the end of intervention (day 2)
  The vignette will be based on hypothetical ex-Boko Haram members, fighter and those forced to join with varying roles within the group and what they did as appropriate. The participants will then be asked 3 sets of outcome measures which relates to Behavioural attitude, emotions and attitude towards reintegration programme.

IPD SHARING:
Plan to Share IPD: No
Data supporting this study cannot be made available due to the sensitive nature and ethical reasons on confidentiality.

REFERENCES:
- [Background] Owonikoko, S. B. (2022). "Take them to government house or Aso Rock": Community receptivity to reintegration of operation safe corridor's deradicalised Ex-Boko Haram members in Northeastern Nigeria. Cogent Social Sciences, 8(1), 2015884.
- [Background] Abdullahi, I., & Onabanjo, H. (2024). Reintegration of ex-combatants and peacebuilding in terrorised communities in northeastern Nigeria. International Journal of Research and Innovation in Social Science (IJRISS), 9 (7), 2283, 2307.